CLINICAL TRIAL: NCT02874417
Title: Computerized Psychoeducation for Anxiety Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Norr01
Record Dates: First submitted 2016-08-08; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Anxiety Sensitivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducation (Experimental): The program was designed to dispel exaggerated thoughts surrounding the danger of the experience of anxiety symptoms, specifically focusing on fears regarding feelings of cognitive dyscontrol. The psychoeducation portion contains video animation and audio narration throughout, as well as some interactive features . Participants are provided with corrective information about the experience of anxiety-related sensations, with a particular focus on dispelling myths commonly held by individuals with high anxiety sensitivity cognitive concerns . Participants are taught that anxiety-related sensations are not dangerous and that they may have developed a conditioned fear to these symptoms of arousal.
  Interventions: Behavioral: CAST psychoeducation
- Health and Wellness (Placebo Comparator): The controlled condition consisted Physical Health Education Training (PHET), a computerized presentation which focuses on information on general healthy living. The PHET program contains information on nutrition, alcohol, water consumption, exercise, sexual health, hygiene, stress management, life organization, social support, positive outlook, and sleep.
  Interventions: Behavioral: PHET

INTERVENTIONS:
Behavioral: CAST psychoeducation
  Arms: Psychoeducation
Behavioral: PHET
  Arms: Health and Wellness

SUMMARY:
This investigation examines the efficacy of a 35 minute computerized psychoeducation protocol in the reduction of elevated anxiety sensitivity cognitive concerns, a risk factor for the development and maintenance of various forms of psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* Elevated Anxiety Sensitivity Cognitive Concerns and indicated by the anxiety sensitivity index-3

Exclusion Criteria:

* History of epilepsy or seizures

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index-3 | 10 minutes post intervention
  Measure of anxiety sensitivity

IPD SHARING:
Plan to Share IPD: Undecided